CLINICAL TRIAL: NCT04515329
Title: Tear Film Markers in Dry Eye Syndrome: Impact of Immunomodulatory Therapy
Brief Title: Tear Film Markers in Dry Eye Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled. Study never started.
Sponsor: Vishal Jhanji (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor-Investigator, Vishal Jhanji, Professor - Cornea Service, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20010206
Record Dates: First submitted 2020-08-05; First posted 2020-08-17 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Cyclosporins; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: * Study arm: Treatment will be commenced with cyclosporine eye drops twice daily with preservative-free artificial tear drops 4 times a day (Treatment).
  * Control arm: Preservative-free artificial tear drops 4 times a day (Control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporine + Artificial Tears (Experimental): Cyclosporine eye drops twice daily (Treatment) with preservative-free artificial tear drops 4 times a day (Control).
  Interventions: Drug: Cyclosporine; Drug: Artificial tear
- Artificial Tears (Other): Preservative-free artificial tear drops 4 times a day (Control).
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Drug: Cyclosporine — Eye drops taken twice daily.
  Other Names: Cequa
  Arms: Cyclosporine + Artificial Tears
Drug: Artificial tear — Preservative-free artificial tear drops 4 times a day.
  Other Names: Preservative-free artificial tears

SUMMARY:
Dry eye is the most common reason for visit to an ophthalmologist's office. The prevalence is on the rise and is mainly attributed to factors such as increased environmental pollution and contact lens use. The current management options are limited to over the counter artificial tear drops and three FDA-approved drugs. Of these, cyclosporine has been used worldwide for treating mild to moderate dry eyes. The earlier version consisted of 0.05% cyclosporine which worked well for a limited number of inflammatory dry eye conditions. Recently, 0.09% cyclosporine was approved by the FDA. The nearly double concentration is expected to be more beneficial for severe inflammation which is often seen in Sjögren syndrome and other Rheumatological conditions associated with dry eyes. In this pilot project, the investigator proposes to evaluate the change in expression of SLURP1 and other markers of ocular surface inflammation before and after treatment with 0.09% cyclosporine eye drops.

DETAILED DESCRIPTION:
Subjects will be recruited based on their diagnosis of dry eyes and an estimate of the severity of the disease that would be made by the investigator based on the patient's history and clinical examination.

Dry Eye Severity is determined by scoring > 12 on the Ocular Surface Disease Index (OSDI) rubric, which is standard practice.

Patients who have been diagnosed with dry eye, but who have not been prescribed a drug to treat that condition, will be recruited.

After signing a consent form, subjects will complete their routine care eye exam.

The PI will include consecutive patients for each arm. Once the mandate is completed in both arms, the investigator will stop the recruitment. The investigator will include patients who will choose to use artificial tear drops in one group. For the other group, the investigator will choose patients who would electively agree to use cyclosporine eyedrops. If these patients choose not to be a part of the study, they will still end up using the treatment that they would like to use.

* Study arm: Treatment will be commenced with cyclosporine eye drops twice daily with preservative-free artificial tear drops 4 times a day (Treatment).
* Control arm: Preservative-free artificial tear drops 4 times a day (Control).

Eye drop timetable:

* If instructed to take 4 times a day, the subject will instill one drop in the morning, the afternoon, the early evening, and before bedtime.
* If instructed to take 2 times a day, the subject will instill one drop in the morning and the evening.
* Subjects will also be instructed to space eye drops by 3-5 minutes.

Both the Cyclosporine and Artificial Tears will be ordered by the subject's doctor, which will be available through the subject's pharmacist. These drops are normally prescribed as part of the subject's routine care.

Both subjects and physicians will be aware of the type of treatment; however the data entry and analysis would be blinded. This will be done by giving each individual subject a linking code.

Subjects will self-administer the eyedrops for 8 weeks.

---------------------------------------------------------

Research Procedures:

The following samples would be collected at baseline and at Week 8:

Baseline (Visit 1):

* Randomization
* Tear Fluid Collection
* Impression Cytology

Week 4 (Visit 2):

• Data collection: Subject will follow up normally with their ophthalmologist as part of their routine care eye exam. The following will be collected: Demographics; Clinical History and office visits; Images and Photography; and Microbiology records.

Week 8 (Visit 3):

* Tear Fluid Collection
* Impression Cytology

Visits 1 and 3 will add up to 20 minutes to the participant's routine care eye exam.

---------------------------------------------------------

Explanation of Procedures:

Numbing Anesthesia Drop (Proparacaine 0.5%):

Subject will receive a numbing anesthesia drop (Proparacaine 0.5%) in the eye that is inflamed as part of their standard of care. The effect of this drop will wear off in 20 minutes after instillation, but the subject is not required to stay until the numbing subsides.

Tear Fluid Collection (Schirmer Testing):

A small amount of the subject's tears will be collected by placing paper strips in the corner of their eye.

Impression Cytology:

The investigators will collect a single sample of material from the surface of the subject's eye and then evaluate it on a cellular level. During impression cytology the subject will be asked to look straight ahead with their chin slightly lifted. A drop of anesthetic eye drops is instilled in the lower fornix of the eye. The plunger of the impression cytology device (EYEPRIM; OPIA Technologies SAS, Paris, France, or equivalent) is pushed to touch the cornea with the membrane gently for 5 seconds. The pressure is released before removing the device. The membrane is then carefully transferred from the device into a 1.5-mL tube using a pair of sterile forceps. Multiple EYEPRIM membranes may be collected. One drop of artificial tear drop would be instilled on the surface of the eye. The participant would be asked to close his/her eye for a few seconds. A capillary tube or Schirmer's strip would be used to collect the tear film.

The total duration of research procedures will be approximately 20 minutes.

---------------------------------------------------------

Samples:

Microbiology analysis will be processed at the UPMC Eye Center's Ophthalmology Microbiology Lab.

The tear fluid samples would be analyzed by ELISA for:

* Matrix metalloproteinase-9
* SLURP-1
* HLA-DR5
* IL-1RA,
* IL-6, and
* IL-8

Impression cytology samples would be used to isolate total RNA, which will be converted to cDNA and used for QPCR evaluation of corresponding transcripts for the above targets. QPCRs along with ELISAs would provide convincing evidence to elucidate the effect(s) of 0.09% cyclosporine on expression of these markers of ocular surface inflammation. At the end of the study, the subject assignments will be unmasked and the difference between the treatment and the control groups analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Dry Eye, but who have not been prescribed a drug to treat this condition.
* 18 years of age and older
* OSDI score > 12

Exclusion Criteria:

* Younger than 18 years of age.
* Any other associated eye diseases other than Dry Eye.
* Inability to understand and give informed consent.
* Patients diagnosed with Dry Eye who are already using Cequa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Tear Film Cytokines | At the time of sample collection (Baseline and Month 6).
  Change from Baseline in tear film cytokines at 6 months. The tear fluid samples would be analyzed by ELISA for: Matrix metalloproteinase-9; SLURP-1; HLA-DR5; IL-1RA; IL-6; and IL-8.

SECONDARY OUTCOMES:
OSDI Score | Last follow-up (Month 6).
  Change is Ocular Surface Disease Index (OSDI) score at Month 6.
  The OSDI quickly assesses the symptoms of ocular irritation in dry eye disease and how they affect functioning related to vision. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Jhanji, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No